CLINICAL TRIAL: NCT05422053
Title: Control-IQ Technology for High Insulin Users With Type 1 Diabetes (Higher-IQ)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tandem Diabetes Care, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TP-0009856
Record Dates: First submitted 2022-06-13; First posted 2022-06-16 (Actual); Results first posted 2024-04-17 (Actual); Last update posted 2025-04-03 (Actual); Status verified 2025-04

CONDITIONS: Type 1 Diabetes
Keywords: Control-IQ; type 1 diabetes; t:slim X2
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- t:slim X2 insulin pump with Control-IQ technology (Experimental): Adults with type 1 diabetes will use the t:slim X2 insulin pump with Control-IQ technology 1.5 for 3-months of outpatient use. Meal and exercise challenges will be performed.
  Interventions: Device: t:slim X2 insulin pump with Control-IQ technology 1.5

INTERVENTIONS:
Device: t:slim X2 insulin pump with Control-IQ technology 1.5 — t:slim X2 insulin pump with Control-IQ technology 1.5, and wearing the Dexcom G6 CGM.

SUMMARY:
A prospective, single-arm study of 13 weeks of home use of the t:slim X2 insulin pump with Control-IQ technology in individuals with type 1 diabetes who will plan to use at least one basal rate > 3 units/hr.

DETAILED DESCRIPTION:
The objectives of the study are to assess safety and explore glycemic outcomes with use of an automated insulin dosing (AID) system (t:slim X2 insulin pump with Control-IQ technology v1.5) in adults with type 1 diabetes who will plan to use at least one basal rate > 3 units/hr. Up to 60 participants may be recruited.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Diagnosis of type 1 diabetes for at least 1 year
* Currently using an insulin pump (of any brand) for at least 3 months, and will plan to use at least one basal rate above 3 units/hr with the study pump
* HbA1c < 10.5%
* Weight ≤ 200 kg
* Residing full-time in the United States, with no anticipated travel outside the United States during the period of study participation.
* Participant has agreed to participate in the study; and has read, understood and signed the informed consent form (ICF); and has agreed to follow all study procedures, including suspending use of any personal CGM for the duration of the clinical trial once the study CGM is in use.
* Willing to use only aspart (novolog) or lispro (humalog) insulin with the study pump, with no use of concentrated insulin above U-100, long-acting basal insulin injections, or inhaled insulin with the study pump.
* Have current glucagon product to treat severe hypoglycemia (injectable or nasal) at home (will provide prescription if they do not have one)
* Willing and able to perform the study exercise and meal challenges.
* Have a care partner, trained in hypoglycemia and hyperglycemia treatment guidelines, present during the challenges and until the next day.
* Investigator has confidence that the participant can successfully operate all study devices and is capable of adhering to the protocol, including ability to respond to alerts and alarms, and to provide basic diabetes self-management.

Exclusion Criteria:

* More than 1 episode of diabetic ketoacidosis (DKA) in the past 6 months
* More than 1 episode of severe hypoglycemia (needing assistance) in the past 6 months
* Inpatient psychiatric treatment in the past 6 months
* History of drug abuse (defined as any illicit drug use) or history of alcohol abuse prior to screening or unwillingness to agree to abstain from illicit drugs throughout the study.
* For Female: Currently pregnant or planning to become pregnant during the time period of study participation
* Use of sulfonylureas, meglitinides or other medications specifically listed in protocol or determined by investigator to interfere with the study
* Unstable dose of SGLT-2 inhibitor, GLP-1 receptor agonist, or DPP-4 inhibitor as listed in the protocol, or starting a new non-insulin glucose lowering or weight loss agent during the trial
* Hemophilia or any other bleeding disorder
* History of heart, liver, lung or kidney disease determined by investigator to interfere with the study
* History of allergic reaction to Humalog or Novolog
* Use of glucocorticoids or other medications determined by investigator to interfere with study
* Abnormal screening electrocardiogram consistent with increased risk during study exercise activities, such as arrhythmia, ischemia, or prolonged QTc interval. Investigator will review all electrocardiograms
* Significant chronic kidney disease (which could impact CGM accuracy in investigator's judgment) or hemodialysis
* History of adrenal insufficiency
* History of abnormal TSH consistent with hypothyroidism or hyperthyroidism that is not appropriately treated
* History of gastroparesis
* A condition, which in the opinion of the investigator or designee, would put the participant or study at risk
* Participation in another pharmaceutical or device trial at the time of enrollment or anticipated for during the time period of study participation
* Employed by, or having immediate family members employed by Tandem Diabetes Care, Inc., or having a direct supervisor at place of employment who is also directly involved in conducting the clinical trial (as a study investigator, coordinator, etc.); or having a first-degree relative who is directly involved in conducting the clinical trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2022-06-29 (Actual); Primary Completion 2023-01-06 (Actual); Study Completion 2023-01-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jordan Pinsker, MD, Study Director — Tandem Diabetes Care
Locations (4):
- United States (4):
  - Barbara Davis Center, Aurora, Colorado
  - Rocky Mountain Diabetes Center, Idaho Falls, Idaho
  - International Diabetes Center, Minneapolis, Minnesota
  - Diabetes & Endocrine Treatment Specialists, Sandy City, Utah

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Carlson AL, Graham TE, Akturk HK, Liljenquist DR, Bergenstal RM, Sulik B, Shah VN, Sulik M, Zhao P, Briggs P, Sassan-Katchalski R, Pinsker JE. Control-IQ Technology Use in Individuals With High Insulin Requirements: Results From the Multicenter Higher-IQ Trial. J Diabetes Sci Technol. 2024 Nov;18(6):1288-1292. doi: 10.1177/19322968241234072. Epub 2024 Mar 5. PMID 38439656

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | t:Slim X2 Insulin Pump With Control-IQ Technology
Started | 34
Completed | 34
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: adults with type 1 diabetes (T1D) who planned to use at least one basal rate > 3 units/hour
Arm/Group | t:Slim X2 Insulin Pump With Control-IQ Technology
Number analyzed (Participants) | 34
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 33
  >=65 years | 1
Age, Continuous [Median (Full Range); unit: years] | 39.9 [20 to 66]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14
  Male | 20
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3
  Not Hispanic or Latino | 31
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 32
  More than one race | 2
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 34
Socio-economic factors (income) [Number; unit: participants]
  Less than $25,000 | 3
  $25,000 to less than $35,000 | 0
  $35,000 to less than $50,000 | 3
  $50,000 to less than $75,000 | 1
  $75,000 to less than $100,000 | 8
  $100,000 to less than $200,000 | 11
  $200,000 or more | 3
  Unknown | 5
Socio-economic factors (education) [Number; unit: participants]
  Less than high school | 1
  High school graduate / diploma / GED | 4
  Some college but no degree | 8
  Associate degree (AA) | 3
  Bachelor's degree (BA, BS, AB) | 13
  Master's degree (MA, MS, MSW, MBA, MPH) | 5
  Professional degree (MD, DDS, DVM, LLB, JD) | 0
  Doctorate degree (PhD, EdD) | 0
  Unknown | 0
  Does not wish to provide | 0
Duration of Diabetes [Mean (Standard Deviation); unit: years] | 21.8 (11.2)
HbA1c at Control-IQ Start [Mean (Standard Deviation); unit: percentage of glycated hemoglobin] | 7.7 (1.1)
BMI [Mean (Standard Deviation); unit: kg/m^2] | 37.6 (5.2)
Total daily insulin [Mean (Standard Deviation); unit: units/kg/day] | 1.2 (0.4)

OUTCOME MEASURES:

1. Primary Outcome: Number of Severe Hypoglycemic Events
Description: Number of severe hypoglycemia events (with cognitive impairment such that assistance of another individual is needed for treatment) during the entire study period
Time Frame: 3 months
Measure: Number; unit: events
Arm/Group | t:Slim X2 Insulin Pump With Control-IQ Technology
Number analyzed (Participants) | 34
events | 0

2. Primary Outcome: Number of Diabetic Ketoacidosis Events
Description: Number of diabetic ketoacidosis events during the entire study period
Time Frame: 3 months
Measure: Number; unit: events
Arm/Group | t:Slim X2 Insulin Pump With Control-IQ Technology
Number analyzed (Participants) | 34
events | 0

3. Primary Outcome: Unanticipated Adverse Device Effects
Description: Number of unanticipated adverse device effects during the entire study period
Time Frame: 3 months
Measure: Number; unit: events
Arm/Group | t:Slim X2 Insulin Pump With Control-IQ Technology
Number analyzed (Participants) | 34
events | 0

4. Primary Outcome: Other Serious Adverse Events
Description: Number of serious adverse events during the entire study period
Time Frame: 3 months
Measure: Number; unit: events
Arm/Group | t:Slim X2 Insulin Pump With Control-IQ Technology
Number analyzed (Participants) | 34
events | 1

5. Secondary Outcome: CGM Time <54 mg/dL Overall
Description: Percent time CGM glucose <54 mg/dL overall
Time Frame: 3 months
Measure: Mean (Standard Deviation); unit: percentage of time
Arm/Group | t:Slim X2 Insulin Pump With Control-IQ Technology
Number analyzed (Participants) | 34
percentage of time | 0.2 (0.2)

6. Secondary Outcome: CGM Time <54 mg/dL Daytime Only
Description: Percent time CGM glucose <54 mg/dL daytime only (06:00 - 24:00)
Time Frame: 3 months
Measure: Mean (Standard Deviation); unit: percentage of time
Arm/Group | t:Slim X2 Insulin Pump With Control-IQ Technology
Number analyzed (Participants) | 34
percentage of time | 0.2 (0.2)

7. Secondary Outcome: CGM Time <54 mg/dL Nighttime Only
Description: Percent time CGM glucose <54 mg/dL nighttime only (00:00 - 06:00)
Time Frame: 3 months
Measure: Mean (Standard Deviation); unit: percentage of time
Arm/Group | t:Slim X2 Insulin Pump With Control-IQ Technology
Number analyzed (Participants) | 34
percentage of time | 0.4 (0.4)

8. Secondary Outcome: CGM Time <70 mg/dL Overall
Description: Percent time CGM glucose <70 mg/dL overall
Time Frame: 3 months
Measure: Mean (Standard Deviation); unit: percentage of time
Arm/Group | t:Slim X2 Insulin Pump With Control-IQ Technology
Number analyzed (Participants) | 34
percentage of time | 1.0 (1.0)

9. Secondary Outcome: CGM Time <70 mg/dL Daytime Only
Description: Percent time CGM glucose <70 mg/dL daytime only (06:00 - 24:00)
Time Frame: 3 months
Measure: Mean (Standard Deviation); unit: percentage of time
Arm/Group | t:Slim X2 Insulin Pump With Control-IQ Technology
Number analyzed (Participants) | 34
percentage of time | 0.9 (0.9)

10. Secondary Outcome: CGM Time <70 mg/dL Nighttime Only
Description: Percent time CGM glucose <70 mg/dL nighttime only (00:00 - 06:00)
Time Frame: 3 months
Measure: Mean (Standard Deviation); unit: percentage of time
Arm/Group | t:Slim X2 Insulin Pump With Control-IQ Technology
Number analyzed (Participants) | 34
percentage of time | 1.4 (1.5)

11. Other Pre Specified Outcome: Hemoglobin A1c
Description: Change in Hemoglobin A1c from baseline
Time Frame: 3 months
Measure: Mean (Standard Deviation); unit: percentage of glycated hemoglobin
Arm/Group | t:Slim X2 Insulin Pump With Control-IQ Technology
Number analyzed (Participants) | 34
percentage of glycated hemoglobin | -0.82 (0.73)
Statistical Analysis 1: Comparison: t:Slim X2 Insulin Pump With Control-IQ Technology; End of Control-IQ Use (13 Weeks) compared to Control-IQ Start; Test type: Superiority; p < 0.001, t-test, 2 sided

12. Other Pre Specified Outcome: CGM Time in Range 70-180 mg/dL Overall
Description: Percent time CGM glucose in range 70-180 mg/dl overall
Time Frame: 3 months
Measure: Mean (Standard Deviation); unit: percentage of time
Arm/Group | t:Slim X2 Insulin Pump With Control-IQ Technology
Number analyzed (Participants) | 34
percentage of time | 64.8 (10.8)

13. Other Pre Specified Outcome: CGM Time in Range 70-180 mg/dL Daytime Only
Description: Percent time CGM glucose in range 70-180 mg/dl daytime only (06:00 - 24:00)
Time Frame: 3 months
Measure: Mean (Standard Deviation); unit: percentage of time
Arm/Group | t:Slim X2 Insulin Pump With Control-IQ Technology
Number analyzed (Participants) | 34
percentage of time | 63.5 (10.9)

14. Other Pre Specified Outcome: CGM Time in Range 70-180 mg/dL Nighttime Only
Description: Percent time CGM glucose in range 70-180 mg/dl nighttime only (00:00 - 06:00)
Time Frame: 3 months
Measure: Mean (Standard Deviation); unit: percentage of time
Arm/Group | t:Slim X2 Insulin Pump With Control-IQ Technology
Number analyzed (Participants) | 34
percentage of time | 68.5 (14.8)

15. Other Pre Specified Outcome: CGM Time >180 mg/dL Overall
Description: Percent time CGM glucose> 180 mg/dL overall
Time Frame: 3 months
Measure: Mean (Standard Deviation); unit: percentage of time
Arm/Group | t:Slim X2 Insulin Pump With Control-IQ Technology
Number analyzed (Participants) | 34
percentage of time | 34.2 (11.1)

16. Other Pre Specified Outcome: CGM Time >180 mg/dL Daytime Only
Description: Percent time CGM glucose> 180 mg/dL daytime only (06:00 - 24:00)
Time Frame: 3 months
Measure: Mean (Standard Deviation); unit: percentage of time
Arm/Group | t:Slim X2 Insulin Pump With Control-IQ Technology
Number analyzed (Participants) | 34
percentage of time | 35.6 (11.3)

17. Other Pre Specified Outcome: CGM Time >180 mg/dL Nighttime Only
Description: Percent time CGM glucose> 180 mg/dL nighttime only (00:00 - 06:00)
Time Frame: 3 months
Measure: Mean (Standard Deviation); unit: percentage of time
Arm/Group | t:Slim X2 Insulin Pump With Control-IQ Technology
Number analyzed (Participants) | 34
percentage of time | 30.1 (15.1)

18. Other Pre Specified Outcome: CGM Time >250 mg/dL Overall
Description: Percent time CGM glucose >250 mg/dL overall
Time Frame: 3 months
Measure: Mean (Standard Deviation); unit: percentage of time
Arm/Group | t:Slim X2 Insulin Pump With Control-IQ Technology
Number analyzed (Participants) | 34
percentage of time | 10.5 (6.8)

19. Other Pre Specified Outcome: CGM Time >250 mg/dL Daytime Only
Description: Percent time CGM glucose >250 mg/dL daytime only (06:00 - 24:00)
Time Frame: 3 months
Measure: Mean (Standard Deviation); unit: percentage of time
Arm/Group | t:Slim X2 Insulin Pump With Control-IQ Technology
Number analyzed (Participants) | 34
percentage of time | 10.7 (6.3)

20. Other Pre Specified Outcome: CGM Time >250 mg/dL Nighttime Only
Description: Percent time CGM glucose >250 mg/dL nighttime only (00:00 - 06:00)
Time Frame: 3 months
Measure: Mean (Standard Deviation); unit: percentage of time
Arm/Group | t:Slim X2 Insulin Pump With Control-IQ Technology
Number analyzed (Participants) | 34
percentage of time | 9.6 (10.4)

21. Other Pre Specified Outcome: CGM Time in Range 70-140 mg/dL Overall
Description: Percent time CGM glucose in range 70-140 mg/dl overall
Time Frame: 3 months
Measure: Mean (Standard Deviation); unit: percentage of time
Arm/Group | t:Slim X2 Insulin Pump With Control-IQ Technology
Number analyzed (Participants) | 34
percentage of time | 37.9 (10.8)

22. Other Pre Specified Outcome: CGM Time in Range 70-140 mg/dL Daytime Only
Description: Percent time CGM glucose in range 70-140 mg/dl daytime only (06:00 - 24:00)
Time Frame: 3 months
Measure: Mean (Standard Deviation); unit: percentage of time
Arm/Group | t:Slim X2 Insulin Pump With Control-IQ Technology
Number analyzed (Participants) | 34
percentage of time | 37.0 (10.8)

23. Other Pre Specified Outcome: CGM Time in Range 70-140 mg/dL Nighttime Only
Description: Percent time CGM glucose in range 70-140 mg/dl nighttime only (00:00 - 06:00)
Time Frame: 3 months
Measure: Mean (Standard Deviation); unit: percentage of time
Arm/Group | t:Slim X2 Insulin Pump With Control-IQ Technology
Number analyzed (Participants) | 34
percentage of time | 40.6 (14.4)

24. Other Pre Specified Outcome: CGM Mean Glucose mg/dL Overall
Description: CGM-measured mean glucose (mg/dL) overall
Time Frame: 3 months
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | t:Slim X2 Insulin Pump With Control-IQ Technology
Number analyzed (Participants) | 34
mg/dL | 167.4 (17.7)

25. Other Pre Specified Outcome: CGM Mean Glucose mg/dL Daytime Only
Description: CGM-measured mean glucose (mg/dL) daytime only (06:00 - 24:00)
Time Frame: 3 months
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | t:Slim X2 Insulin Pump With Control-IQ Technology
Number analyzed (Participants) | 34
mg/dL | 168.8 (17.3)

26. Other Pre Specified Outcome: CGM Mean Glucose mg/dL Nighttime Only
Description: CGM-measured mean glucose (mg/dL) nighttime only (00:00 - 06:00)
Time Frame: 3 months
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | t:Slim X2 Insulin Pump With Control-IQ Technology
Number analyzed (Participants) | 34
mg/dL | 163.1 (25.1)

27. Other Pre Specified Outcome: Coefficient of Variation Overall
Description: CGM measured glucose variability measured with the coefficient of variation overall
Time Frame: 3 months
Measure: Mean (Standard Deviation); unit: percentage of coefficient of variation
Arm/Group | t:Slim X2 Insulin Pump With Control-IQ Technology
Number analyzed (Participants) | 34
percentage of coefficient of variation | 34.7 (5.1)

28. Other Pre Specified Outcome: Coefficient of Variation Daytime Only
Description: CGM measured glucose variability measured with the coefficient of variation daytime only (06:00 - 24:00)
Time Frame: 3 months
Measure: Mean (Standard Deviation); unit: percentage of coefficient of variation
Arm/Group | t:Slim X2 Insulin Pump With Control-IQ Technology
Number analyzed (Participants) | 34
percentage of coefficient of variation | 34.4 (4.6)

29. Other Pre Specified Outcome: Coefficient of Variation Nighttime Only
Description: CGM measured glucose variability measured with the coefficient of variation nighttime only (00:00 - 06:00)
Time Frame: 3 months
Measure: Mean (Standard Deviation); unit: percentage of coefficient of variation
Arm/Group | t:Slim X2 Insulin Pump With Control-IQ Technology
Number analyzed (Participants) | 34
percentage of coefficient of variation | 33.7 (6.4)

30. Other Pre Specified Outcome: Standard Deviation of Glucose, Overall
Description: CGM measured standard deviation of glucose (mg/dL) overall
Time Frame: 3 months
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | t:Slim X2 Insulin Pump With Control-IQ Technology
Number analyzed (Participants) | 34
mg/dL | 58.2 (11.7)

31. Other Pre Specified Outcome: Standard Deviation of Glucose, Daytime
Description: CGM measured standard deviation of glucose (mg/dL), daytime only (06:00 - 24:00)
Time Frame: 3 months
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | t:Slim X2 Insulin Pump With Control-IQ Technology
Number analyzed (Participants) | 34
mg/dL | 58.4 (11.0)

32. Other Pre Specified Outcome: Standard Deviation of Glucose, Nighttime Only
Description: CGM measured standard deviation of glucose (mg/dL), nighttime only (00:00 - 06:00)
Time Frame: 3 months
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | t:Slim X2 Insulin Pump With Control-IQ Technology
Number analyzed (Participants) | 34
mg/dL | 55.1 (14.3)

ADVERSE EVENTS:
Time Frame: 13 weeks
Arm/Group | t:Slim X2 Insulin Pump With Control-IQ Technology
All-Cause Mortality (participants affected / at risk) | 0/34
Serious Adverse Events (participants affected / at risk) | 1/34
Other Adverse Events (participants affected / at risk) | 19/34
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | t:Slim X2 Insulin Pump With Control-IQ Technology (N=34)
New onset atrial fibrillation (Cardiac disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | t:Slim X2 Insulin Pump With Control-IQ Technology (N=34)
Otitis media (Ear and labyrinth disorders) | 1 (1)
Tympanic membrane perforation (Ear and labyrinth disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1)
Tooth fracture (Gastrointestinal disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1)
Influenza like illness (General disorders) | 1 (1)
Bronchitis (Infections and infestations) | 1 (1)
COVID-19 (Infections and infestations) | 2 (2)
Ear Infection (Infections and infestations) | 1 (1)
Influenza (Infections and infestations) | 2 (2)
Otitis Externa (Infections and infestations) | 1 (1)
Pharyngitis streptococcal (Infections and infestations) | 1 (1)
Tooth abscess (Infections and infestations) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 7 (10)
Skin abrasion (Injury, poisoning and procedural complications) | 1 (1)
Ketonemia (Metabolism and nutrition disorders) | 1 (1)
Dyslipidemia (Metabolism and nutrition disorders) | 1 (1)
Ligament sprain (Musculoskeletal and connective tissue disorders) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1)
Stiff person syndrome (Musculoskeletal and connective tissue disorders) | 1 (1)
Migraine (Nervous system disorders) | 1 (1)
Chronic kidney disease (Renal and urinary disorders) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Sleep apnea syndrome (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Hypertension (Vascular disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-03-21): https://cdn.clinicaltrials.gov/large-docs/53/NCT05422053/Prot_SAP_000.pdf